CLINICAL TRIAL: NCT05413005
Title: A Randomized, Open-label, Pilot Study Evaluating the Efficacy of Extracorporeal Photopheresis (ECP) in the Treatment of Type 1 Diabetes Mellitus
Brief Title: Efficacy of Extracorporeal Photopheresis (ECP) in the Treatment of Type 1 Diabetes Mellitus
Acronym: OPERA
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abu Dhabi Stem Cells Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT.004.1.1.OPERA
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Extracorporeal photopheresis; ECP
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Photopheresis; Therapeutics

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated (1:1) in a parallel assignment involving two groups of participants: Group A (Regular-intensity arm): ECP on a regular-intensity regimen described in the Protocol as add-on T1DM standard of care, or Group B (Accelerated-intensity arm): ECP on an accelerated regimen plus T1DM standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (ECP regular-intensity arm) (Experimental): ECP in a regular-intensity arm plus T1DM standard of care
  Interventions: Combination Product: ECP regular-intensity arm; Biological: T1DM standard of care
- Group B (ECP accelerated-intensity arm) (Experimental): ECP in an accelerated-intensity arm plus T1DM standard of care
  Interventions: Combination Product: ECP accelerated-intensity arm; Biological: T1DM standard of care

INTERVENTIONS:
Combination Product: ECP regular-intensity arm — * Weeks 1-8: Once every 2 weeks: weeks 1, 3, 5, 7 (cryo-ECP bags infused twice-a-week)
  * Weeks 9-16: Once per month: weeks 9, 13 (cryo-ECP bags infused once-a-week)
  * Weeks 17-24: One: week 17 (cryo-ECP bags infused every two weeks)
  Other Names: Extracorporeal photochemotherapy; Extracorporeal photoimmunotherapy
  Arms: Group A (ECP regular-intensity arm)
Combination Product: ECP accelerated-intensity arm — * Weeks 1-8: Once every week: weeks 1- 7 (cryo-ECP bags infused twice-a-week)
  * Weeks 9-16: Cryo-ECP bags infused once-a-week
  * Weeks 17-24: Cryo-ECP bags infused every two weeks
  Other Names: Extracorporeal photochemotherapy; Extracorporeal photoimmunotherapy
  Arms: Group B (ECP accelerated-intensity arm)
Biological: T1DM standard of care — The standard of care is defined as per the "DOH Standards for diagnosis, management and data reporting for diabetes" in combination with the DOH recommended NICE guidelines "Type 1 diabetes in adults: diagnosis and management (NG17)"
  Other Names: Multiple Dose Injection (MDI) therapy

SUMMARY:
OPERA Study is a randomized, open-label, prospective, pilot, and a monocentric clinical trial involving outpatients within Abu Dhabi Stem Cells Center (ADSCC) with a confirmed diagnosis of type 1 diabetes mellitus (T1DM). The patients will be randomly allocated (1:1) in a parallel assignment involving two groups of participants: Group A (Regular-intensity arm): Extracorporeal Photopheresis (ECP) on a regular-intensity regimen described in the Protocol as add-on T1DM standard of care, or Group B (Accelerated-intensity arm): ECP on an accelerated regimen plus T1DM standard of care.

DETAILED DESCRIPTION:
The standard of care is defined as per the "DOH Standards for diagnosis, management and data reporting for diabetes" in combination with the DOH recommended NICE (UK National Institute for Health and Care Excellence) guidelines "Type 1 diabetes in adults: diagnosis and management (NG17)". OPERA Study will be fully conducted in ADSCC, including the patient assessment and inclusion, randomization, ECP procedures, and follow-up consultations, according to this Protocol and GCP principles. All patients will receive T1DM standard of care, plus additional ECP protocols on two regimens of investigational interventions. The primary objective is the safety assessment of ECP, to be assessed by the tolerability to the ECP procedures, incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) assessed by the CTCAE v5.0, and the WHO-UMC causality assessment system. The other primary objective is the preliminary efficacy assessment of the ECP as an add-on treatment to the standard of care for T1DM patients, assessed by the exogenous insulin use, HbA1c levels, C-peptide levels, and clinically important hypoglycemic episodes. The secondary objective is the assessment of the immune response profile in T1DM patients receiving standard of care and additional ECP procedures. The trial is approved by the institutional ADSCC Research Ethics Committee (REC) and written informed consent will be obtained from all patients. OPERA Study will be conducted following the principles of the Declaration of Helsinki and ICH-GCP guidelines.

ELIGIBILITY:
* Inclusion Criteria

  * Confirmed and documented diagnosis of T1DM. Patients must have:
  * A documented history of T1DM within the first 3 years of onset.
  * Should be on a multiple dose injection (MDI) therapy.
  * C-Peptide levels of ˂ 0.7 ng/mL.
  * HbA1C ≥ 6.5% to ≤ 10%.
  * Evidence of pancreatic autoimmunity, if available (positive anti-glutamic acid decarboxylase [GAD]; Islet antigen 2 [anti-IA2]; and/or zinc transporter 8 [ZnT8] antibodies).
  * Male or female aged ≥ 18 to ≤ 50 years.
  * Weight > 40 kg.
  * Hematocrit ≥ 32%.
  * Platelet count ≥ 100 x10^9/L (with or without transfusion support).
  * Willingness to participate in all OPERA Study tests, visits, and ECP procedures, as outlined in the informed consent.
  * Willingness to use at least one reliable method of birth control (e.g. abstinence, oral contraceptives, intrauterine devices, barrier method with spermicide, or surgical sterilization) throughout the study for all men and women of childbearing potential.
  * The patient agrees to participate in the trial, and signs the OPERA Study informed consent form.
* Exclusion Criteria

  * Pediatric aged < 18 or ˃ 50 years.
  * Clinical diagnosis of type 2 diabetes mellitus (T2DM).
  * Inability to tolerate fluid changes associated with ECP (e.g. inadequate renal, hepatic, pulmonary and cardiac function leading to enable patient to tolerate extracorporeal volume shifts associated with ECP).
  * Hypersensitivity or allergy to citrate products.
  * Hypersensitivity or allergy to psoralen compounds such as Methoxsalen (8-Methoxypsoralen, 8-MOP).
  * Aphakia (8-MOP is contraindicated because of the significantly increased risk of retinal damage due to the absence of lenses).
  * Presence of comorbidities that may result in photosensitivity (systemic lupus erythematosus, porphyries, albinism, etc.).
  * Suspected or diagnosed Diabetic Ketoacidosis (DKA) at the moment of the screening visit.
  * Uncontrolled infection requiring treatment at study entry.
  * Laboratory evidence of any of the following:
  * White Blood Cell (WBC) count < 3.00 x10^9/L.
  * Serum transaminase levels > x2 upper normal limit (UNL).
  * Hematocrit < 32%.
  * Platelet count < 100 x10^9/L (with or without transfusion support).
  * Diagnostic of Hepatitis B Virus (HBV) infection.
  * Diagnostic of Human Immunodeficiency Virus (HIV) infection or Acquired Immunodeficiency Syndrome (AIDS).
  * Pregnant or lactating women.
  * Have participated in other clinical trial in the past 3 months.
  * Organ transplants in the past 3 months.
  * Current diagnosis of cancer.
  * Inability to comply with all OPERA Study tests, visits, and procedures (including ECP).
  * Inability to provide informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability to ECP procedures | Weeks 0 - 24
  Rate of tolerability of the ECP will be assessed by the number of ECP discontinuation due to adverse events (AE), or withdrawal of participants of the Study due to serious adverse events (SAEs)
Incidence of adverse events (AEs) | Weeks 0 - 24
  Incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs): Proportion of participants with AEs as assessed by CTCAE v5.0
Exogenous insulin use | Baseline, months 3, 6, and 12
  Rate of modification in exogenous insulin requirements compared with baseline. Marker for efficacy of treatment: reducing insulin dose
HbA1c levels | Baseline, months 3, 6, and 12
  Rate of modification in HbA1c levels compared with baseline. Marker for efficacy of treatment: decreasing for a target HbA1c level of 48 mmol/mol [6.5%]
C-peptide levels | Baseline, months 3, 6, and 12
  Rate of modification in C-Peptide levels compared with baseline. Marker for efficacy of treatment: increasing C-Peptide levels of ≥ 0.7 ng/mL
Clinically important hypoglycemic episodes | Baseline - Month 12
  Frequency of clinically important hypoglycemic episodes (described in Protocol).
  Marker for efficacy of treatment: requiring decrease of insulin dose)

SECONDARY OUTCOMES:
Immune response profile (cellular) | Baseline, months 3, 6, and 12
  CD3, CD4, CD8, CD11c, CD14, CD16, CD19, CD20, CD25, CD27, CD28, CD38, CD45, CD45RA, CD45RO, CD56, CD57, CD66b, CD123, CD127, CD161, CD294, CCR4, CCR6, CCR7, CXCR3, CXCR5, will be assessed for identification of immune cells and subsets analyses
Serum IgG levels | Baseline, months 3, 6, and 12
  Serum IgG concentration will be assessed for characterization of the humoral response profile
Serum IgA levels | Baseline, months 3, 6, and 12
  Serum IgA concentration will be assessed for characterization of the humoral response profile
Serum IgM levels | Baseline, months 3, 6, and 12
  Serum IgM concentration will be assessed for characterization of the humoral response profile

CONTACTS AND LOCATIONS:
Overall Officials: Yandy M Castillo-Aleman, MD, Principal Investigator — Abu Dhabi Stem Cells Center
Locations (1):
- Abu Dhabi Stem Cells Center, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No